CLINICAL TRIAL: NCT05653882
Title: An Open-Label Phase 1a/1b Dose-Escalation and Expansion Study Investigating the Safety, Pharmacokinetics, Pharmacodynamics, and Activity of AB248 Alone or in Combination With Pembrolizumab in Adult Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study Evaluating AB248 Alone or in Combination With Pembrolizumab in Adult Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Asher Biotherapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB248-101; KEYNOTE-E29 (Other: Merck Sharp & Dohme LLC); MK-3475-E29 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer; Melanoma; Squamous Cell Carcinoma of Head and Neck; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- etakafusp alfa (AB248) Monotherapy Dose-Escalation (Experimental): etakafusp alfa (AB248) will be administered intravenously as a single agent
  Interventions: Biological: etakafusp alfa (AB248)
- etakafusp alfa (AB248) + pembrolizumab Combination Dose-Escalation (Experimental): etakafusp alfa (AB248) and pembrolizumab will be administered intravenously
  Interventions: Biological: etakafusp alfa (AB248); Biological: pembrolizumab
- etakafusp alfa (AB248) Monotherapy Indication Expansion (Experimental): etakafusp alfa (AB248) will be administered intravenously as a single agent in disease specific cohorts
  Interventions: Biological: etakafusp alfa (AB248)
- etakafusp alfa (AB248) + pembrolizumab Combination Indication Expansion (Experimental): etakafusp alfa (AB248) and pembrolizumab will be administered intravenously in disease specific cohorts
  Interventions: Biological: etakafusp alfa (AB248); Biological: pembrolizumab

INTERVENTIONS:
Biological: etakafusp alfa (AB248) — Intravenous infusion of etakafusp alfa (AB248): CD8+ T cell selective interleukin-2 investigational drug
Biological: pembrolizumab — Intravenous infusion of pembrolizumab
  Other Names: KEYTRUDA®
  Arms: etakafusp alfa (AB248) + pembrolizumab Combination Dose-Escalation; etakafusp alfa (AB248) + pembrolizumab Combination Indication Expansion

SUMMARY:
This is a phase I, First-in-Human (FIH), open-label study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and preliminary efficacy of AB248 as monotherapy OR in combination with pembrolizumab in adult participants with locally advanced or metastatic solid tumors. The study will consist of a dose escalation and a dose expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age at the time consent is signed.
* Has adequate end organ function per laboratory testing.
* Pregnancy prevention requirements
* Has measurable disease per RECIST 1.1 as assessed by the local site Investigator/radiology.
* Has a performance status of 0 or 1 on Eastern Cooperative Oncology Group scale.
* Histologic documentation of incurable, locally advanced or metastatic tumor of the type being evaluated in individual cohorts

Exclusion Criteria:

* Has a diagnosis of immunodeficiency.
* Has a history of a previous, additional malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has an active infection requiring systemic therapy.
* Inability to comply with study and follow-up procedures.
* Has had a severe hypersensitivity reaction (Grade ≥3) to treatment with pembrolizumab, another monoclonal antibody, or has history of any hypersensitivity to any components of the study treatments or any of their excipients.
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks (or, if shorter, within 5 half-lives for kinase inhibitors) prior to first dose of study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment or has had a history of radiation pneumonitis.
* Receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.
* Has received previous treatment with another agent targeting the IL-2, IL-7, or IL-15 receptors.
* Is expected to require any other form of antineoplastic therapy while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Dose-Limiting Toxicities (DLTs) | From Study Day 1 through up to Day 21, Day 28, or Day 42
  Based on toxicities observed
Frequency of Serious Adverse Events (SAEs) | Signed consent up to 90 days after discontinuing study treatment
  Based on toxicities observed
Frequency of Treatment Emergent Adverse Events (TEAEs) | Study Day 1 up to 90 days after discontinuing study treatment
  Based on toxicities observed
Frequency of Adverse Events of Special Interest (AESIs) | Study Day 1 up to 90 days after discontinuing study treatment
  Based on toxicities observed
Frequency of Adverse Events (AEs) leading to dose interruption or treatment discontinuation and death | Signed consent up to 90 days after discontinuing study treatment
  Based on toxicities observed

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as the proportion of subjects with confirmed complete response (CR) or partial response (PR); a confirmed response is a response that persists on repeat-imaging ≥4 weeks after initial documentation of response.
Duration of Response (DOR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as time from date of first objective response (either CR or PR) to first documentation of radiographic disease progression.
Disease Control Rate (DCR) according to RECIST version 1.1 | Study Day 1 up to approximately 24 months
  Defined as the percentage of patients who have achieved CR, PR, or stable disease.
Progression-Free Survival (PFS) according to RECIST version 1.1 | Study Day 1 until the date of first documented progression or date of death from any cause, assessed up to approximately 24 months
  Defined as the time from first dose of AB248 to first documentation of radiographic disease progression or death, whichever occurs first
Overall Survival (OS) according to RECIST version 1.1 | Study Day 1 up to time of death, assessed up to approximately 24 months
  Defined as the time from first dose of AB248 to the date of death.
Maximum observed blood concentration (Cmax) of AB248 | Study Day 1 up to approximately 24 months
  Defined as assessments for measuring maximum blood concentration of AB248
AUC Area under the Plasma Concentration versus Time Curve (AUC) of AB248 | Study Day 1 up to approximately 24 months
  Defined as assessments for evaluating the Area Under the Concentration-Time Curve (AUC)
Elimination half-life (t1/2) of AB248 | Study Day 1 up to approximately 24 months
  Defined as the time required for half of the drug to be eliminated from the blood
Quantification of peripheral blood CD8+ T cell pharmacodynamics | Study Day 1 up to approximately 24 months
  Defined as the volumetric enumeration of CD8+ T cells in whole blood as assessed by flow cytometry
Changes in CD8+ T cell density in tumor tissues | Study Day 1 to approximately 1 month
  Defined as changes in immune-staining for CD8+ T cells density in tumor tissue from patients providing paired biopsies.
Frequency of anti-drug antibodies (ADA)s to AB248 | Study Day 1 up to approximately 24 months
  Defined as the frequency of ADA formation for immunogenicity assessments evaluated during study treatment up until 30 days after the final dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Asher Biotherapeutics, Inc.
Locations (20):
- United States (20):
  - City of Hope, Duarte, California
  - UCLA, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California
  - Yale, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Rutgers, New Brunswick, New Jersey
  - NYU, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Intermountain Health, Murray, Utah
  - Virginia Commonwealth, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No